CLINICAL TRIAL: NCT03856918
Title: Optimal Level of Positive End-expiratory Pressure to Reduce Postoperative Atelectasis After Lung Resection With Protective One-lung Ventilation
Brief Title: Optimal Level of PEEP in Protective One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-1901-086-1004
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Video-assisted Thoracic Surgery; Postoperative Atelectasis; Positive End-expiratory Pressure
Keywords: Protective ventilation; One-lung ventilation
MeSH Terms: interventions — Positive-Pressure Respiration; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEEP 3 cm of water (Experimental): Patients allocated in this group will be applied protective one-lung ventilation using tidal volume of 5 ml/kg predicted body weight with PEEP of 3 cm of water during thoracic surgery.
  Interventions: Procedure: PEEP 3 cm of water
- PEEP 6 cm of water (Experimental): Patients allocated in this group will be applied protective one-lung ventilation using tidal volume of 5 ml/kg predicted body weight with PEEP of 6 cm of water during thoracic surgery.
  Interventions: Procedure: PEEP 6 cm of water
- PEEP 9 cm of water (Experimental): Patients allocated in this group will be applied protective one-lung ventilation using tidal volume of 5 ml/kg predicted body weight with PEEP of 9 cm of water during thoracic surgery.
  Interventions: Procedure: PEEP 9 cm of water

INTERVENTIONS:
Procedure: PEEP 3 cm of water — PEEP of 3 cm of water will be applied during one-lung ventilation.
  Arms: PEEP 3 cm of water
Procedure: PEEP 6 cm of water — PEEP of 6 cm of water will be applied during one-lung ventilation.
  Arms: PEEP 6 cm of water
Procedure: PEEP 9 cm of water — PEEP of 9 cm of water will be applied during one-lung ventilation.
  Arms: PEEP 9 cm of water

SUMMARY:
Protective ventilation strategy has been widely applied in the field of thoracic surgery requiring one-lung ventilation to reduce postoperative pulmonary complications. Low tidal volume, positive end-expiratory pressure (PEEP), and intermittent recruitment maneuver are key components of protective ventilation strategy. Recent evidence suggests that a tidal volume of 4-5 ml/kg should be applied during protective one-lung ventilation. However, optimal level of PEEP is still unclear. This study aims to investigate optimal level of PEEP to minimize postoperative atelectasis by comparing modified lung ultrasound score in patients applied protective one-lung ventilation using PEEP of 3, 6, or 9 cm of water during thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Video-assisted Thoracic Surgery under one-lung ventilation

Exclusion Criteria:

* Moderate to severe obstructive/restrictive pattern in preoperative pulmonary function test
* Chronic kidney disease
* Coronary artery disease
* Pulmonary hypertension
* Bilateral lung surgery
* Conversion to thoracotomy
* American Society of Anesthesiologists physical status IV or more
* Refusal to participate

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Modified lung ultrasound score | Postoperative 1 hour
  The score is calculated by adding up the 12 individual quadrant scores assessed using lung ultrasound.

SECONDARY OUTCOMES:
Intraoperative desaturation | Average time of 60-90 minutes
  Oxygen saturation by pulse oximetry <95% during one-lung ventilation
Intraoperative partial pressure of arterial oxygen/fraction of inspired oxygen ratio | Average time of 60-90 minutes
  partial pressure of arterial oxygen/fraction of inspired oxygen ratio during one-lung ventilation
Postoperative desaturation | Postoperative 24 hours
  Oxygen saturation by pulse oximetry <95%
plasma Tumor Necrosis Factor-α | 10 minutes after initiation of one-lung ventilation
  proinflammatory cytokine
plasma Interleukin-6 | 10 minutes after initiation of one-lung ventilation
  proinflammatory cytokine
plasma Interleukin-10 | 10 minutes after initiation of one-lung ventilation
  anti-inflammatory cytokine
Postoperative pulmonary complication | Postoperative 7 days
  Composite outcome of atelectasis, pneumonia, acute respiratory distress syndrome, or pulmonary aspiration

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Hyon Bahk, MD,PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea